CLINICAL TRIAL: NCT05699031
Title: The PROTECT-study: Home-based Telerehabilitation in the Post-operative Care After Shoulder Arthroplasty Compared to Usual Care: a Randomized Control Trial
Brief Title: Shoulder Prosthesis Telerehab Care Trial
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2022-0357
Record Dates: First submitted 2022-12-23; First posted 2023-01-26 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: SHOULDER ARTHROPLASTY; REHABILITATION; TELEREHABILITATION
Keywords: SHOULDER ARTHROPLASTY; REHABILITATION; TELEREHABILITATION
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP-GROUP (Experimental): Patients allocated in the app-group will use the app to rehabilitate.
  Interventions: Device: APP
- PHYSIO-GROUP (Active Comparator): Patients allocated in the physio-group will rehabilitate according to the usual care protocol
  Interventions: Other: PHYSICAL THERAPY

INTERVENTIONS:
Device: APP — Patients allocated in the app-group will use the newly developed smartphone app te rehabilitate. 5 exercises are provided daily. Daily questionnaires will monitor exercise performance, VAS pain, household activities. Information modules will be sent at specific times.
  Arms: APP-GROUP
Other: PHYSICAL THERAPY — Patients allocated in the physio-group will go, twice a week, to a physical therapist of their choice to rehabilitate. The physical therapist will follow the general guidelines provided by the hospital (surgeon).
  Other Names: PHYSIO-GROUP
  Arms: PHYSIO-GROUP

SUMMARY:
The goal of this clinical trial is to compare the rehabilitation by use of a smartphone-app with the usual care of physical therapy in patients, 60 years and older, who underwent a primary shoulder arthroplasty.

The main questions it aims to answer are:

* is the outcome of rehabilitation with the app as good as the usual care?
* is the outcome for both types of shoulder arthroplasty similar?
* what is the usability of the app?.

Participants will

* have treatment according to the group they are allocated to
* fill in questionnaires at specific moments during the rehabilitation stage (0 - 3 months ) and at 1 year post-surgery

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* primary total shoulder arthroplasty (anatomical and reverse)
* osteoarthritis, cuff tear arthropathy, pseudoparalysis
* return home after discharge from hospital
* no brace after surgery
* sufficient verbal and written comprehension
* hospitalization insurance

Exclusion Criteria:

* revision arthroplasty
* arthroplasty for fracture or tumor
* neurological disease (parkinson, stroke, ...)
* no access to smartphone, tablet or internet connectivity

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
SHOULDER PAIN AND DISABILITY INDEX (SPADI)_baseline pre-operative | Prior to surgery
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
SHOULDER PAIN AND DISABILITY INDEX (SPADI)_baseline post-operative | week 0
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | week 3
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | week 6
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | week 12
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | week 52
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder

SECONDARY OUTCOMES:
ACTIVE MOBILITY (ROM) OF THE SHOULDER | Prior to surgery, week 3, week 6, week 12, week 52
  ACTIVE ROM: forward flexion and abduction with extended elbow, functional internal and external rotation in standing position.
  * maximal pain free ROM
  * forward flexion and abduction with extended elbow: measured with the EasyAngle (Meloq AB Sweden)
  * hand-to-back and hand-nek test : scored as in Constant-Murley Score
    2) PASSIVE: forward flexion, abduction, external and internal rotation in supine position.
  * maximal pain free ROM
  * forward flexion and abduction: measured with the EasyAngle (Meloq AB Sweden)
  * rotations: measured as ER1 (arm at the side)/ ER2 (arm in 90° abduction) and IR1 (arm in 90° forward flexion)/ IR2 (arm in 90° abduction) with the EasyAngle (Meloq AB Sweden).
PASSIVE MOBILITY (ROM) OF THE SHOULDER | Prior to surgery, week 3, week 6, week 12, week 52
  PASSIVE: forward flexion, abduction, external and internal rotation in supine position.
  * maximal pain free ROM
  * forward flexion and abduction: measured with the EasyAngle (Meloq AB Sweden)
  * rotations: measured as ER1 (arm at the side)/ ER2 (arm in 90° abduction) and IR1 (arm in 90° forward flexion)/ IR2 (arm in 90° abduction) with the EasyAngle (Meloq AB Sweden).
STRENGTH | Prior to surgery, week 3, week 6, week 12, week 52
  Forward flexion, extension, ab- and adduction, external and internal rotation.
  * isometrical contraction for 5 seconds, 3 repetitions, 30 sec break in between
  * measured with EasyForce (Meloq AB Sweden)
  * seated, both feet on the ground, back against backrest
  * elbow flexed (90°) held at side, fist forward, thumb upward
CONSTANT-MURLEY SCORE | Prior to surgery, week 3, week 6, week 12, week 52
  Content: partially clinical (65 points) and partially PROM (35 points) assessed.
  Scoring: The formula to calculate the total score is:" pain (0-15) + ADL (4x (0-5) = 0-20) + mobility (4 x (0-10) = 0-40) + strength (0 -25)". Strength will be measured with the arm elevated to 90 ° in the scapular plane using an IDOmeter.
  Interpretation: 0-55 points = bad, 56-70 points = mediocre, 71-85 points = good, 86-100 points = excellent score
ACTIVITIES OF DAILY LIVING EXTERNAL AND INTERNAL ROTATIONS (ADLEIR) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 12 questions about specific ADL tasks that require external or internal rotation while performing.
  Scoring: Each activity is scored between 0 (unable to do) and 3 (not difficult at all). All activities should be performed without the help of flexing the neck or bending the trunk and without the help of first abducting the elbow (i.e., without doing a hornblower sign).
  Interpretation: The maximal score is 36. A higher score means that the patient is able to perform ADL activities with enough strength in external and internal rotation
SINGLE ASSESSMENT NUMERIC EVALUATION (SANE) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 1 question: 'how would you rate your shoulder today as a percentage of normal?'.
  Scoring: percentage between 0 and 100% Interpretation: 100% being a normal shoulder.
EUROQOL 5-DIMENSIONS 5-LEVEL (EQ-5D-5L) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 5 questions + EQ-5D VAS for general health. Scoring: 5-response scale (from 'no problems' to 'extreme problems') + VAS percentage between 0 (worst imaginable health state) and 100 (best imaginable health state).
  Interpretation: VAS score for general health indicates how a patient perceives his general health, Other questions are descriptive for problems in mobility, self-care, usual activities, pain/ discomfort, anxiety/depression.
GRONINGEN ACTIVITY RESTRICTION SCALE (GARS-4) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 18 questions to identify problems with self-sufficiency in self-care and housekeeping. Patients do not respond if they do that activity but rather if they could do that activity.
  Scoring: ordinal scale from 1 (Yes, I can do that on my own without any effort) up to 4 (No, I can't do that on my own, but only with the help of others).
  Interpretation: A higher score (max 72) is related to a lower self-sufficiency.
EXERCISE ADHERENCE RATING SCALE (EARS) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 3 sections section A: 6 questions to evaluate the prescribed exercises. section B: 6 questions on how a patient does the recommended exercises or activities.
  section C: 10 statements on why a patient does or does not do the recommended exercises or activities.
  Scoring: sections B and C: 5-point Likert scale (0 - 4) (some questions scored reversed).
  Interpretation:
  section B (range 0 - 24): a higher score indicates a better compliance/adherence .
  section C (range 0 - 40): a higher score indicates a better adherence.
EXERCISE DIARY | Daily post-surgery (week 0 - week 12)
  Content: performed exercises, household activities, VAS pain. Diary on paper for physio-group, by the app for the app-group.
SELF-EFFICACY FOR EXERCISES (SEE) | Week 3, week 6, week 12, week 52
  Content: 9 questions about 'confidence in engaging in exercise 3 times a week for 20 minutes if faced with a barrier'.
  Scoring: 'not very confident' (0) and 'very confident' (10). Interpretation: The higher the score , the patient feel more confident in performing prescribed exercises.
GLOBAL RATING OF CHANGE SCALE (GROC) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: A single question (How would you currently describe the change in your operated shoulder compared to just before surgery) is scored on a scale, ranging from 'very much worse' through 'unchanged' to 'completely recovered'.
  Scoring: The scale used is divided in 11 points ( very much worse -5, the same 0, very much better + 5) Interpretation: the number given indicates how a patient perceives the change after surgery.
GLOBAL PERCEIVED EFFECT (GPE/GEE) | Prior to surgery, week 3, week 6, week 12, week 52
  Content: 2 questions: To what extent have you recovered from your symptoms?, How satisfied are you with your treatment?.
  Scoring: a 7-point rating scale. Interpretation: The higher the score , the better.

OTHER OUTCOMES:
M-HEALTH APP USABILITY QUESTIONNAIRE (MAUQ) | Week 12
  Content: 21 questions in 3 categories: ease of use and satisfaction, system information arrangement, usefulness (version for interactive app, user patient and provider).
  Scoring: between 1 (strongly disagree) and 7 (strongly agree) => average score. Interpretation: the higher the score the higher the usability.
SYSTEM USABILITY SCALE (SUS) | Week 12
  Content: 10 questions about system satisfaction, usability and learnability. Scoring: 5 response options ranging from strongly disagree (1) to strongly agree (5).
  Interpretation: A score above 68 (/100) is considered above average, while a score lower than 68 is considered a below average score.
SINGLE EASE QUESTION (SEQ) | Week 12
  Content: 1 question to assess how difficult users find a task. Scoring: 7-point rating scale ranging from very difficult (1) to very easy (7).
  Interpretation: The average SEQ score is 5.5 (between 5.3 and 5.6). It is advised to ask a more detailed information/ explanation if a score <5 is given.
AGE | Pre-surgery
  Content: specify age of participant
GENDER | Pre-surgery
  Content: specify gender of participant
DIAGNOSTICS | Pre-surgery
  Content: specify why patient needed a shoulder arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Van Tongel, PhD, Principal Investigator — University Ghent, University Hospital Ghent; Ann Cools, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No